CLINICAL TRIAL: NCT02630303
Title: Phase I Study of High Fluence Light Emitting Diode-Red Light (LED-RL) in Human Skin
Brief Title: High Fluence Light Emitting Diode-Red Light (LED-RL) in Human Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jared Jagdeo, MD, MS (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency); East Bay Institute for Research and Education (Other)
Responsible Party: Sponsor-Investigator, Jared Jagdeo, MD, MS, Medical Physician, VA Northern California Health Care System
Organization: VA Northern California Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-12-00756
Record Dates: First submitted 2015-12-09; First posted 2015-12-15 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Fibrosis; Scarring; Scar; Wounds; Injuries; Keloid; Cicatrix; Hypertrophic
Keywords: light emitting diode-red light; LED-RL; high fluence; skin fibrosis; wound healing; scar; keloid; RCT
MeSH Terms: conditions — Fibrosis; Cicatrix; Wounds and Injuries; Keloid; Hypertrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LED-RL Phototherapy (Experimental): The protocol for dose escalation requires subjects be enrolled sequentially in groups of five (three subjects randomized to LED-RL phototherapy and two subjects randomized to mock therapy).
  After either a maximally tolerated dose (MTD) has been established, or the study endpoint of 640 J/cm2 has been achieved, an additional 27 LED-RL phototherapy subjects (for a total of 30) and 18 mock therapy subjects (for a total of 20) (determined randomly) will be enrolled to satisfy Hanley's Rule of Three, such that it can be concluded with 95% confidence that fewer than 1 person in 10 will experience an adverse event.
  Interventions: Device: LED-RL Phototherapy
- Mock Therapy (Sham Comparator): The protocol for dose escalation requires subjects be enrolled sequentially in groups of five (three subjects randomized to LED-RL phototherapy and two subjects randomized to mock therapy).
  After either a maximally tolerated dose (MTD) has been established, or the study endpoint of 640 J/cm2 has been achieved, an additional 27 LED-RL phototherapy subjects (for a total of 30) and 18 mock therapy subjects (for a total of 20) (determined randomly) will be enrolled to satisfy Hanley's Rule of Three, such that it can be concluded with 95% confidence that fewer than 1 person in 10 will experience an adverse event.
  Interventions: Device: Mock Therapy

INTERVENTIONS:
Device: LED-RL Phototherapy — The maximum recommended starting dose (MSRD) (160 J/cm2) will be administered to Group 1's LED-RL phototherapy randomized subjects and the LED-RL dose will be escalated in subsequent groups using the classical method for dose escalation as described by Spilker: starting with dose (X) increased by an equal amount (in this instance: X=160 J/cm2, 2X=320 J/cm2, 3X=480 J/cm2, 4X=640 J/cm2). Common expected procedure side effects are mild and temporary, including warmth, redness (erythema) and swelling (edema). The maximally tolerated dose (MTD) is defined as the dose level below the dose producing unacceptable but reversible toxicity and is considered the upper limit of subject tolerance.
  All subjects will receive total of nine LED-RL phototherapy, three times per week for three consecutive weeks.
  Other Names: Omnilux New-U (Photo Therapeutics, Carlsbad, CA)
  Arms: LED-RL Phototherapy
Device: Mock Therapy — Mock therapy will be administered to mock therapy randomized subjects using the mock therapy unit and only generates warmth and does not emit LED-RL.
  All subjects will receive total of nine mock therapy procedures, three times per week for three consecutive weeks.
  Other Names: Mock therapy unit (Photo Therapeutics, Carlsbad, CA)
  Arms: Mock Therapy

SUMMARY:
The goal of this study is to establish the safety of high fluence LED-RL from 160 J/cm2 up to 640 J/cm2 in healthy subjects. The hypothesis is that high fluence LED-RL phototherapy is safe in human skin.

DETAILED DESCRIPTION:
Skin fibrosis is involved in a variety of pathologic processes ranging from exuberant scar formation secondary to surgery or trauma, as in hypertrophic and keloid scars, to immune-mediated processes such as scleroderma and chronic graft-versus-host disease. As highlighted by quality-of-life studies, skin fibrosis imparts a significant socioeconomic burden due to the functional, aesthetic, and psychosocial impact it has on a patient's life. The effects of visible light, while common in the environment (visible spectrum accounts for 44% of total solar energy), remain undefined. An important safety feature of visible red light (600 nm to 700 nm) is that it does not generate pro-carcinogenic DNA damage as does ultraviolet (UV) light. Recently published clinical observations indicate that red light in combination with other modalities such as photosensitizers in combined red light photodynamic therapy can lessen skin fibrosis. However, preliminary in vitro data generated by the investigator's research group suggests that red light can function as a stand-alone treatment, eliminating the side-effects of chemical photosensitizers and the potential long-term harm of current UV therapy. Furthermore, commercially available light emitting diode-red light (LED-RL) units exist and are already FDA-cleared for other dermatological uses (such as rhytides and acne), thus clinical translation for use in skin fibrosis could occur relatively quickly following safety and efficacy demonstration. Developing high fluence LED-RL phototherapy as a treatment for skin fibrosis would represent an important advance in scarring conditions that lacks the serious systemic side effects associated with immunomodulatory agents (such as oral steroids); avoids the need for invasive, painful injections with anti-fibrotic agents (such as intralesional steroids, 5-fluorouracil and bleomycin); and eliminates the UV-induced DNA damage associated with skin cancer and photoaging that are associated with current UVA/UVA1 and UVB/narrowband UVB phototherapy. To the investigator research group's knowledge, no clinical trials have been performed to determine the safety of high fluence LED-RL for treatment of skin fibrosis. Therefore, the innovation of this approach is that the investigator research group intend to study high fluence LED-RL as a safe modality for treatment of skin fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of any sex, ethnicity and age
* Nondominant proximal anterior forearm is wide enough to ensure reproducible placement of LED-RL phototherapy or mock therapy hand-held unit
* Available and willing to attend all clinic visits
* Able and willing to give informed consent

Exclusion Criteria:

* Subjects using any photosensitizers (i.e. lithium, melatonin, phenothiazine antipsychotics, antibiotics)
* Subjects with diabetes mellitus (DM)
* Subjects with a history of skin cancer; basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
* Subjects with systemic lupus erythematous (SLE)
* Subjects with any other medical condition that could be compromised by exposure to the proposed treatment
* Subjects with light-sensitive conditions or on photosensitizing medications (All subjects will be tested for photosensitivity per manufacturer user guide instructions)
* Subjects with open wounds on the nondominant proximal anterior forearm
* Subjects with fibrotic skin disease or other skin conditions on the nondominant proximal anterior forearm
* Subjects with tattoos that cover the procedure site on the nondominant proximal anterior forearm

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incidence of procedure-related common expected procedure outcomes and adverse events (safety and tolerability) | 3 weeks
  To evaluate safety of high fluence LED-RL Phototherapy by recording any common expected procedure outcomes [warmth, erythema (redness), and edema (swelling) that are mild, self-limited, and are expected to last less than 24 hours] and adverse events (including: second-degree or higher skin burning or blistering, erythema lasting more than 24 hours, severe swelling, pain, ulceration, change in sensation, and/or muscle weakness], via assessment during and immediately post-procedure, subject diary of adverse events and weekly phone calls)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD, MS, Principal Investigator — Sacramento VA Medical Center- Dermatology Service
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

REFERENCES:
- [Result] Jagdeo JR, Adams LE, Brody NI, Siegel DM. Transcranial red and near infrared light transmission in a cadaveric model. PLoS One. 2012;7(10):e47460. doi: 10.1371/journal.pone.0047460. Epub 2012 Oct 15. PMID 23077622
- [Result] Mamalis A, Jagdeo J. Light-emitting diode-generated red light inhibits keloid fibroblast proliferation. Dermatol Surg. 2015 Jan;41(1):35-9. doi: 10.1097/01.DSS.0000452650.06765.51. PMID 25485805
- [Result] Sadick NS. A study to determine the efficacy of a novel handheld light-emitting diode device in the treatment of photoaged skin. J Cosmet Dermatol. 2008 Dec;7(4):263-7. doi: 10.1111/j.1473-2165.2008.00404.x. PMID 19146602
- [Result] Sadick NS. Handheld LED array device in the treatment of acne vulgaris. J Drugs Dermatol. 2008 Apr;7(4):347-50. PMID 18459515
- [Result] Lev-Tov H, Mamalis A, Brody N, Siegel D, Jagdeo J. Inhibition of fibroblast proliferation in vitro using red light-emitting diodes. Dermatol Surg. 2013 Aug;39(8):1167-70. doi: 10.1111/dsu.12212. Epub 2013 Apr 16. PMID 23590233
- [Derived] Ho D, Kraeva E, Wun T, Isseroff RR, Jagdeo J. A single-blind, dose escalation, phase I study of high-fluence light-emitting diode-red light (LED-RL) on human skin: study protocol for a randomized controlled trial. Trials. 2016 Aug 2;17:385. doi: 10.1186/s13063-016-1518-7. PMID 27484782